CLINICAL TRIAL: NCT01242397
Title: Prospective.Randomized, Blinded, Crossover Chronic IDE Study of the Effects of Pacing on Mitral Regurgitation in Patients Without Standard Indications for Cardiac Resynchronization Therapy
Brief Title: Mitral Insufficiency Reduction With Biventricular Pacing
Acronym: MiRBi
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Trinity Medical Center, Illinois (Other)
Collaborators: Medtronic (Industry); Duke University (Other); Massachusetts General Hospital (Other); Augusta University (Other)
Responsible Party: Helbert Acosta MD, Trinity Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MiRBi- Acosta
Record Dates: First submitted 2010-11-10; First posted 2010-11-17 (Estimated); Last update posted 2010-12-02 (Estimated); Status verified 2009-11

CONDITIONS: Mitral Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CRT ON (Other): After implant, patients will be randomized to CRT pacing ON vs OFF in crossover fashion with 3 months in each period
  Interventions: Device: CRT pacing
- CRT- OFF (Other): After implant, patients will be randomized to CRT pacing OFF vs ON in crossover fashion with 3 months in each period
  Interventions: Device: CRT pacing

INTERVENTIONS:
Device: CRT pacing — The chronic effect of CRT pacing on the degree of MR in pts with severe-to-moderate or severe functional MR. The treatment being studied is CRT pacing therapy with standard of care LV lead placement. Patients will be randomized to CRT pacing ON vs. OFF and followed for a total of up to 8 months. This includes two 3-month crossover periods for each pacing modality (CRT ON and CRT OFF) and a 6-week washout period between these periods.

SUMMARY:
The purpose of this study is to show that CRT(Cardiac Resynchronization Therapy) pacing in patients with severe functional MR (Mitral Regurgitation) who are not currently indicated for CRT will demonstrate chronic benefit of MR reduction( via echo measured MR/LA area and ERO per American Society of ECHO guidelines) and to show that CRT pacing is safe in these patients.

DETAILED DESCRIPTION:
Approximately 50 patients will be randomized, followed and analyzed in this prospective study. Patients who meet all inclusion and no exclusion criteria will be enrolled and implanted with a CRT system. Baseline evaluation, which includes clinical symptom evaluation and an echocardiogram, will be performed at the time of randomization, which should occur as soon after device implant as possible but no later than 2 week post -implant. The baseline echocardiogram should be acquired prior to the device being programmed to the randomized setting. Repeat echocardiograms and scheduled follow-up evaluations will be performed at the end of each 3 month crossover period.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age
* Patients with moderate-to-severe or severe functional MR.

  * EROA > 40 mm2 and an MR/LA > 40% (severe)
  * 30 ≤ EROA ≤ 40 mm2 and 30 ≤ MR/LA ≤ 40% (moderate-to-severe)
* Baseline rates of 50-90 beats per minute (patients with sinus rhythm) or AF
* QRS < 120 ms
* LVEF < 35%
* Willing to sign informed consent
* On standard stable heart failure medical regimen (beta blockers and ACE-I or ARBs) for at least 1 month before randomization, if tolerated
* Patient has the ability to understand the requirements of the study, including consent for use and disclosure of research-related information
* Patient has the ability to comply with study procedures and protocol, including required study visits

Exclusion Criteria:

* candidate for CRT or has a previously implanted CRT device
* previously implanted implantable pulse generators (IPG) or implantable cardioverter defibrillator (ICD) with at least 10 % pacing in the right ventricle
* patient has life expectancy <6 months
* patient is pregnant
* significant aortic stenosis
* uncontrolled hypertension
* mitral valve stenosis
* severe mitral valve calcification
* ruptured chordae tendinae or papillary muscle
* mitral valve leaflet disorders (i.e. endocarditis, lupus, tumors, rheumatic heart disease)
* chronic mitral leaflet degeneration (ie. Marfans)
* previous valve replacement or surgery
* IV inotropes or IV vasodilators
* candidate for mitral valve repair or replacement surgery within the next 6 months
* patient has in-hospital acute coronary syndrome (ACS) (NSTEMI/STEMI) prior to randomization
* patient has planned or elective percutaneous coronary intervention (PCI) or other non-cardiac surgery prior to randomization
* patient is currently enrolled in an investigational drug or device study
* patient is clinically unstable per PI assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Chronic(8 months post-implant) benefit of MR reduction | Chronic
  To show that CRT pacing in patients with severe functional MR who are not currently indicated for CRT will demonstrate chronic(8 months post-implant) benefit of MR reduction (via echo measured MR/LA area and ERO per American Society of Echo guidelines)

SECONDARY OUTCOMES:
To compare MR Severity (ERO and MR/LA area), heart volume and dimensions via echo and clinical symptoms between two pacing modalities | Chronic
  Secondary objectives will compare MR severity (ERO and MR/LA area), heart volume and dimensions via echo (LA and LV), LVEF via echo (Simpson's method and clinical sypmtoms (NYHA class, QOL, 6MHW distance) between the two pacing modalities (CRT ON and OFF)

CONTACTS AND LOCATIONS:
Overall Officials: Helbert Acosta, MD, Principal Investigator — Trinity Medical Center; Patrick Hranitzky, MD, Principal Investigator — Duke University; Jagmeet Singh, MD, Principal Investigator — Massachusetts General Hospital; Adam A Berman, MD, Principal Investigator — Augusta University